CLINICAL TRIAL: NCT02762409
Title: Improve the Quality of Life After a Hospitalization in Critical Care Thanks to a Program of Prevention of Discomforts Perceived by the Patients of Critical Care Base on Targeted Measures
Brief Title: Improve the Quality of Life After a Hospitalization in Critical Care
Acronym: AQVAR
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier of Chartres (Other)
Responsible Party: Sponsor
Other Study IDs: PREPS-15-15-0183
Record Dates: First submitted 2016-04-18; First posted 2016-05-05 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2016-08

CONDITIONS: Depression; Depression Symptoms
Keywords: critical care; reduction of depression syndrome; anxiety; quality of life; post traumatic stress; discomforts
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: None Retained — The calculation of the number of necessary subjects is realized from the main criterion and bases on the proportion of presenting subjects of the clinically significant depressive symptoms in 1 year of their hospitalization in intensive care, estimated from it under scale D of the score HAD-S.The proposal of the subject waited for the patient presenting this profile was on the works available in particular on the general review of DAVYDOW and AL
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- patients exposed: Patients exposed will be estimated in the study IPREA3 corresponding to surviving individuals of a hospitalization in intensive care in a department having set up the program of reduction of the discomforts collected by the patients of intensive care during a minimal period of 5 months. The program is so defined as factor of exposure and supposed protector of development of anxio-depressive disorders.These patients will have been included in the study IPREA3 in 17 centers of the interventional group of the study IPREA3 during the months of April, 2015 and October, 2015, and in 17 centers of the group control some study IPREA3 during October 2015
  Interventions: Other: experimental
- patients non exposed: The patients "not exposed" in the supposed factor protector of development of anxio-depressive disorders will be constituted by the patients estimated in the study IPREA3 corresponding to surviving individuals of a hospitalization in intensive care in a department having never operated the program of reduction of the discomforts collected by the patients of intensive care. These patients will have been included in the study IPREA3 in 17 centers of the group control some study IPREA3 during October 2014 and April, 2015 and in 17 centers of the interventional group during October 2014
  Interventions: Other: control

INTERVENTIONS:
Other: experimental — corresponding to surviving individuals of a hospitalization in intensive care in a department having set up the program of reduction of the discomforts collected by the patients of intensive care during a minimal period of 5 months. The program is so defined as factor of exposure and supposed protector of development of anxio-depressive disorders.These patients will have been included in the study IPREA3 in 17 centers of the interventional group of the study IPREA3 during the months of April, 2015 and October, 2015
  Groups: patients exposed
Other: control — The patients "not exposed" in the supposed factor protector of development of anxio-depressive disorders will be constituted by the patients estimated in the study IPREA3 corresponding to surviving individuals of a hospitalization in intensive care in a department having never operated the program of reduction of the discomforts collected by the patients of intensive care. These patients will have been included in the study IPREA3 in 17 centers of the group control some study IPREA3 during October 2014 and April, 2015
  Groups: patients non exposed

SUMMARY:
Demonstrate that the IPREA3 program (Study: Impact of Multicomponent Intervention to Reduce Perceived Discomforts of the patients in intensive care) reducing discomforts perceived by the patients of intensive care, implemented at the level of the whole intensive care unit, reduce the incidence of the depressive symptoms one year after intensive care exit.

DETAILED DESCRIPTION:
AQVAR is a study of type not exposed presentations, study ancillary of controlled study, multicentric with randomization to cluster, the study IPREA3, for which a financing was already obtained within the framework of the Hospital National Clinical Program of Research on 2012, current study, the inclusions of which began on October 1st, 2014 after the obtaining of all the necessary authorizations. To date, more than 4300 patients were included in the study IPREA3 within 34 departments or intensive care units participating on approval. All the patients included in the study AQVAR will be patients included before in the study IPREA3 and which a complete questionnaire IPREA3 of measure of the discomforts collected by all the patients of intensive care will be available.

The AQVAR study leans on the original current research IPREA3 which consists of the evaluation of a program with multiple components of reduction of the discomforts collected by the patients of including in intensive care:

1. The preliminary identification of a binomial doctor-nurse of local coordinating experts of the program IPREA3
2. A systematic measure of the discomforts collected by means of the questionnaire IPREA administered the day of the exit.
3. An immediate return of the scores of discomfort in every nursing administering the questionnaire IPREA
4. The implementation of measures targeted by reduction of the discomforts, based on the analysis of the results appropriate to the intensive care unit.

The innovative character is also brought by the research for the association between conditions of hospitalization in intensive care according to the perception of the patient and very remote quality of life of the hospitalization in intensive care , as well as by the evaluation of a method of primary prevention of the psychiatric morbidity post-intensive care.

The individual profits waited for the patient hospitalized in an intensive care unit having implemented the program of reduction of the discomforts IPREA3 are the improvement of its conditions of hospitalization during its whole stay in intensive care, such as the patient perceives them at the exit of intensive care, then remote, a reduction of the risk of arisen a state of post-traumatic stress, anxious and/or depressive symptoms, and cognitive dysfunctions. This reduction of the psychiatric morbidity should lead to an improvement of its quality of life bound to the health, but also to the recourse to the consultations in an emergency department or to the new hospitalizations.

The expected main collective profits are a better description of the post-traumatic states of stress consecutive to a hospitalization in intensive care, as well as an understanding of mechanisms and risk factors of arisen this psychiatric morbidity.

If the study AQVAR allows to show the tested hypothesis, it will be an additional, decisive argument, to implement in all the intensive care units a program with multiple components of type IPREA3 of reduction of the received discomforts, requiring the commitment of all the healthcare professionals, whose feasibility is in the course of demonstration, and which must be integrated into the projects of department and establishment.

The additional expected collective profits concern two other populations:

* The close relations of the patients hospitalized in intensive care, according to the hypothesis of an interaction between the quality of life of the patients after the intensive care and that of their susceptible close relations they too to develop a state of post-traumatic stress after the hospitalization in intensive care.
* The health workers practicing in intensive care, among which the job satisfaction, and possibly the level risks of professional exhaustion, should be improved by the membership in a department applying the program, federative, of reduction of the discomforts in intensive care, applied by the whole team specialized in intensive care.

ELIGIBILITY:
Inclusion Criteria:

The same criteria of the IPREA3 study

* Taken out alive of intensive care
* Hospitalization in intensive care extending at least over three calendar days.

Exclusion Criteria:

* Deaths in intensive care
* Age 18-year-old inferior
* Under guardianship patient
* Incompatible situation with the administration of the IPREA questionnaire at the exit of intensive care: presence of neuropsychic disorders, language barrier, transfer under mechanical ventilation, taken out of intensive care in urgency
* Patient refused to participate in the study IPREA3
* Patient refused to participate in the study AQVAR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients included in the study AQVAR will be patients included before in the study IPREA3 for whom the IPREA3 questionnary of measure of the discomforts collected by the patients will be informed (available score for each of the items establishing the questionnaire IPREA3). The inclusion of the patients in the study AQVAR will be made the day of the intensive care exit.
Sampling Method: Non-Probability Sample
Enrollment: 1006 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Improve the reduction of depressive symptoms | up to 52 weeks of the hospitalization
  A score 8 (maximal score of 21) allows to hold the presence of clinically significant depressive symptoms.

SECONDARY OUTCOMES:
Score of the sub-scale A of the questionnaire HAD-S ( Hospital and Anxiety Depression Scale) | up to 52 weeks of the hospitalization
  Allowing to estimate the presence of anxious symptoms. Score of the sub-scale A of the questionnaire HAD-S one year after the exit of intensive care allowing to estimate the presence of anxious symptoms. A score 8 (maximal score of 21) allows to hold the presence of clinically significant anxious symptoms.
  The scale HAD contains 14 highly-rated items from 0 to 3. Seven questions relate to the anxiety ( total A) and seven others in the depressive dimension (total D), so allowing the obtaining of two scores, the maximal note of wich for each of them is 21.
Score IES-R ( impact of Events Scale-Revised) | up to 52 weeks of the hospitalization
  Allowing to detect a risk of state of post traumatic stress.
Questionnaire EQ-5D | up to 52 weeks of the hospitalization
  Indicators of quality of life estimated by questionnaires EQ-5D
Describe quality of life | up to 52 weeks of the hospitalization
  Return home, taken by a professional activity, an existence of a psychiatric or psychological follow up, and a regular consumption of psychotropics
Duration of hospitalization | Consecutive to the hospitalization in intensive care
  Informations are in the medical bases statistic of each hospital

CONTACTS AND LOCATIONS:
Overall Officials: Pierre KALFON, PhD, Principal Investigator — CH CHARTRES
Locations (12):
- France (12):
  - C.H. de Chartres, Chartres
  - CHU Beaujon APHP, Clichy
  - CH Douai, Douai
  - CH La Rochelle, La Rochelle
  - CH Le Puy en Velay, Le Puy-en-Velay
  - CH Lens, Lens
  - CHU Edouard Herriot, Lyon
  - CHU Saint Louis APHP, Paris
  - CHU Cochin APHP, Paris
  - CHU NHC, Strasbourg
  - CHU Hautepierre, Strasbourg
  - CH Troyes, Troyes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Griffiths J, Fortune G, Barber V, Young JD. The prevalence of post traumatic stress disorder in survivors of ICU treatment: a systematic review. Intensive Care Med. 2007 Sep;33(9):1506-18. doi: 10.1007/s00134-007-0730-z. Epub 2007 Jun 9. PMID 17558490
- [Result] Pandharipande PP, Girard TD, Ely EW. Long-term cognitive impairment after critical illness. N Engl J Med. 2014 Jan 9;370(2):185-6. doi: 10.1056/NEJMc1313886. No abstract available. PMID 24401069
- [Result] Davydow DS, Hough CL, Zatzick D, Katon WJ. Psychiatric symptoms and acute care service utilization over the course of the year following medical-surgical ICU admission: a longitudinal investigation*. Crit Care Med. 2014 Dec;42(12):2473-81. doi: 10.1097/CCM.0000000000000527. PMID 25083985
- [Result] Davydow DS, Zatzick D, Hough CL, Katon WJ. A longitudinal investigation of posttraumatic stress and depressive symptoms over the course of the year following medical-surgical intensive care unit admission. Gen Hosp Psychiatry. 2013 May-Jun;35(3):226-32. doi: 10.1016/j.genhosppsych.2012.12.005. Epub 2013 Jan 28. PMID 23369507
- [Result] Kalfon P, Mimoz O, Auquier P, Loundou A, Gauzit R, Lepape A, Laurens J, Garrigues B, Pottecher T, Malledant Y. Development and validation of a questionnaire for quantitative assessment of perceived discomforts in critically ill patients. Intensive Care Med. 2010 Oct;36(10):1751-1758. doi: 10.1007/s00134-010-1902-9. Epub 2010 May 26. PMID 20502874
- [Derived] Kalfon P, Alessandrini M, Boucekine M, Renoult S, Geantot MA, Deparis-Dusautois S, Berric A, Collange O, Floccard B, Mimoz O, Julien A, Robert R, Audibert J, Renault A, Follin A, Thevenin D, Revel N, Venot M, Patrigeon RG, Signouret T, Fromentin M, Sharshar T, Vigne C, Pottecher J, Levrat Q, Sossou A, Garrouste-Orgeas M, Quenot JP, Boulle C, Azoulay E, Baumstarck K, Auquier P; IPREA-AQVAR Study Group. Tailored multicomponent program for discomfort reduction in critically ill patients may decrease post-traumatic stress disorder in general ICU survivors at 1 year. Intensive Care Med. 2019 Feb;45(2):223-235. doi: 10.1007/s00134-018-05511-y. Epub 2019 Jan 30. PMID 30701294